CLINICAL TRIAL: NCT02125760
Title: The RETORNUS Study: Dual Training to Restore the Function of Respiratory Muscles in Stroke Patients
Brief Title: Respiratory Muscle Training in Subacute Stroke Patients
Acronym: RETORNUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Esther Marco Navarro, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSM/RHB/NR/14; RETORNUS (Other: PSMAR)
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Muscle Weakness
Keywords: Respiratory muscle training; stroke; rehabilitation
MeSH Terms: conditions — Muscle Weakness; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiratory Muscle Training (IMT) (Sham Comparator): Patients with subacute stroke in a neurorehabilitation setting.
  Interventions: Other: Inspiratory Muscle Training (IMT)
- High-intensity IMT (Experimental): Patients with subacute stroke in a neurorehabilitation setting.
  Interventions: Other: High-intensity IMT

INTERVENTIONS:
Other: Inspiratory Muscle Training (IMT) — Sham IMT at a fixed workload of 10 cmH2O. 5 sets of 10 repetitions, twice a day, 7 days per week, for 4 weeks.
  Other Names: No applicable
  Arms: Inspiratory Muscle Training (IMT)
Other: High-intensity IMT — High Intensity IMT. The training load is the maximum inspiratory load defined according to patient tolerance. This load will be equivalent to 10 maximal repetitions (RM) as 10 consecutive inspirations (x 5 sessions), twice a day.
  Other Names: Short duration respiratory muscle training
  Arms: High-intensity IMT

SUMMARY:
This study is divided for development in two complementary work packages justified by the need to incorporate new strategies to optimize rehabilitation outcomes in stroke patients. The general objectives are: 1) to determine the prevalence of respiratory muscle dysfunction in stroke patients; 2) to identify the existence of a potential amino acid marker of increased risk of muscle dysfunction after suffering a stroke; 3) to evaluate the effectiveness of incorporating the respiratory muscle training as an innovative adjuvant therapy in stroke rehabilitation program that may decrease the incidence of morbidity and mortality in the medium and long term; and 4) to quantify the potential impact of respiratory muscle training on the costs of care for stroke patients.

DETAILED DESCRIPTION:
Stroke is a major cause of morbidity and mortality worldwide. It determines a substantial socioeconomic burden. Stroke can lead to varying degrees of oropharyngeal dysphagia (25-85% of patients) and respiratory muscle dysfunction associated with an increase in medical complications such as bronchoaspiration pneumonia, malnutrition and death. The respiratory muscle dysfunction is a common functional abnormality in chronic respiratory diseases such as chronic obstructive pulmonary disease (COPD), heart failure, multiple sclerosis in which it has been shown to modify the expected survival. Dysphagia is present in a significant proportion of patients admitted to Rehabilitation (up to 85% depending on series) in the subacute phase of stroke. There is no drug able to restore the swallowing function and inspiratory and expiratory muscle function in these patients. Consequently, neurological rehabilitation is the mainstay of treatment of these disorders.

Amino acids (AA) are essential for proper protein synthesis. Skeletal muscle represents the largest reserve of body AA, which may be used according to metabolic needs. Within this group of compounds, the most involved in muscle metabolism are glutamate, aspartate, asparagine, valine, leucine and isoleucine. A pathobiological association between decrease in muscle glutamate and diaphragm dysfunction in patients with chronic respiratory diseases has been demonstrated in chronic respiratory patients. Moreover, glutamate levels of the diaphragm can be restored as a result of muscle training, playing a decisive role as a precursor of certain AA (glutamine and alanine), and glutathione in patients with COPD. Other studies have defined that glutamine may be a biomarker of training response in healthy individuals. Several publications have reflected the decrease of glutamine and glutamate as a result of different diseases and in some cases have tried to supplement this deficit.

Muscle dysfunction is defined as a function impairment (decrease in strength and/or resistance) of muscles whose main consequence is muscle fatigue. Although exercise training has been used successfully to restore function in patients with some chronic illnesses and frailty, there is little evidence of the beneficial effects of an overall muscle training in stroke patients. Regarding peripheral muscles, a high-intensity training improves strength and endurance of lower limbs muscles (paretic and non paretic) in stroke patients. Dysfunction of the diaphragm and other respiratory muscles has important clinical implications. It associates with susceptibility to hypercapnic ventilatory failure, ineffective cough, and even higher incidence of repeated hospital admissions and mortality. Therefore, respiratory muscle weakness described in some stroke patients justifies the need to train respiratory muscles because there is no general exercise (bicycle, legs, arms) able to induce an overload enough to achieve training effect on respiratory muscles.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegia secondary to first ischemic stroke in the subacute phase, and
* informed consent signed by the candidates of the study, after receiving full information on objectives, techniques and possible consequences.

Exclusion Criteria:

* Serious cardiovascular, neuromuscular or metabolic conditions that could interfere with the results and/or interfere with the measurements,
* significant alcohol abuse (> 80 g/day) or severe malnutrition, and
* treatment with drugs with potential effect on muscle structure and function (steroids, anabolic steroids, thyroid hormones and immunosuppressants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | 3 weeks
  Respiratory muscle strength is assessed through maximal inspiratory and expiratory pressures (MIP and MEP, respectively) using a pressure transducer connected to a digital register system. The MIP is measured at mouth during a maximum effort from residual volume against occluded airway. To determine the MEP, the patients will perform a maximum expiratory effort from total lung capacity (TLC) in the face of the occluded airway. A specific and validated respiratory pressures manometer will be used (Micro RPM, Cardinalhealth, Kent, UK). For the purposes of the study, 'responders' will include the group of patients with an increase of 25% or more in respiratory muscle strength (MIP and MEP).
  Measures will be done once every week

SECONDARY OUTCOMES:
Handgrip strength assessment | 3 weeks
  Handgrip strength will be assessed during maximal voluntary isometric contraction of the flexor muscles of the fingers, using a dynamometer (JAMAR, Nottinghamshire, UK). We consider both the non-dominant and dominant hand. Reference values are those from Webb et al. (J Par Ent Nutr 1989, 13:30-3).
  Measures once every week
Lower limb strength measurement | 3 weeks
  Lower limb strength will be measured during a maximal voluntary isometric knee extension while the patient is sit in a bank of exercise (DOMYOS HG 050, Decathlon, France). An isometric dynamometer Nicholas Manual Muscle Tester (NMMT) (Lafayette Instrument Company, Lafayette, Indiana) will be used according to Dunn JC (J Phys Ther Ger 2003).
  Measures once every week
Serum aminoacids analysis | Up to 3 weeks
  Analysis of plasma samples (high performance liquid chromatography (HPLC) will determine levels of glutamine, valine, isoleucine, leucine and glutamate at baseline and at the end of muscle training using the technique previously described and validated (Clin Chem 1988, 34 (12): 2510-3). Venous blood samples will be collected in heparinized tube and centrifuged to obtain plasma. Later proceed to deproteinization with sulfosalicylic acid for analyzing the concentration of amino acids (AA). Finally the sample will be frozen at -80 º C for further analysis.
Adverse events as a measure of safety and tolerability | 18 months after discharge
  Comorbidity variables (occurrence of complications, hospital admissions, hospital length of stay) and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Duarte, MD, PhD, Study Director — Institut Hospital del Mar d'Investigacions Mèdiques. Universitat Autònoma de Barcelona.
Locations (1):
- Physical Medicine and Rehabilitation Dpt. Parc de Salut Mar, Hospital del Mar, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Kumar S, Selim MH, Caplan LR. Medical complications after stroke. Lancet Neurol. 2010 Jan;9(1):105-18. doi: 10.1016/S1474-4422(09)70266-2. PMID 20083041
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Teixeira-Salmela LF, Parreira VF, Britto RR, Brant TC, Inacio EP, Alcantara TO, Carvalho IF. Respiratory pressures and thoracoabdominal motion in community-dwelling chronic stroke survivors. Arch Phys Med Rehabil. 2005 Oct;86(10):1974-8. doi: 10.1016/j.apmr.2005.03.035. PMID 16213241
- [Background] Terre R, Mearin F. Oropharyngeal dysphagia after the acute phase of stroke: predictors of aspiration. Neurogastroenterol Motil. 2006 Mar;18(3):200-5. doi: 10.1111/j.1365-2982.2005.00729.x. PMID 16487410
- [Background] Indredavik B, Rohweder G, Naalsund E, Lydersen S. Medical complications in a comprehensive stroke unit and an early supported discharge service. Stroke. 2008 Feb;39(2):414-20. doi: 10.1161/STROKEAHA.107.489294. Epub 2007 Dec 20. PMID 18096834
- [Background] Martin BJ, Corlew MM, Wood H, Olson D, Golopol LA, Wingo M, Kirmani N. The association of swallowing dysfunction and aspiration pneumonia. Dysphagia. 1994 Winter;9(1):1-6. doi: 10.1007/BF00262751. PMID 8131418
- [Background] Schmidt J, Holas M, Halvorson K, Reding M. Videofluoroscopic evidence of aspiration predicts pneumonia and death but not dehydration following stroke. Dysphagia. 1994 Winter;9(1):7-11. doi: 10.1007/BF00262752. PMID 8131429
- [Background] Dall'Ago P, Chiappa GR, Guths H, Stein R, Ribeiro JP. Inspiratory muscle training in patients with heart failure and inspiratory muscle weakness: a randomized trial. J Am Coll Cardiol. 2006 Feb 21;47(4):757-63. doi: 10.1016/j.jacc.2005.09.052. Epub 2006 Jan 26. PMID 16487841
- [Background] Chiara T, Martin AD, Davenport PW, Bolser DC. Expiratory muscle strength training in persons with multiple sclerosis having mild to moderate disability: effect on maximal expiratory pressure, pulmonary function, and maximal voluntary cough. Arch Phys Med Rehabil. 2006 Apr;87(4):468-73. doi: 10.1016/j.apmr.2005.12.035. PMID 16571384
- [Background] Logemann JA. Treatment of oral and pharyngeal dysphagia. Phys Med Rehabil Clin N Am. 2008 Nov;19(4):803-16, ix. doi: 10.1016/j.pmr.2008.06.003. PMID 18940642
- [Background] Carnaby G, Hankey GJ, Pizzi J. Behavioural intervention for dysphagia in acute stroke: a randomised controlled trial. Lancet Neurol. 2006 Jan;5(1):31-7. doi: 10.1016/S1474-4422(05)70252-0. PMID 16361020
- [Background] Wheeler KM, Chiara T, Sapienza CM. Surface electromyographic activity of the submental muscles during swallow and expiratory pressure threshold training tasks. Dysphagia. 2007 Apr;22(2):108-16. doi: 10.1007/s00455-006-9061-4. Epub 2007 Feb 10. PMID 17294298
- [Background] Huckabee ML, Doeltgen S. Emerging modalities in dysphagia rehabilitation: neuromuscular electrical stimulation. N Z Med J. 2007 Oct 12;120(1263):U2744. PMID 17972964
- [Background] Shaw GY, Sechtem PR, Searl J, Keller K, Rawi TA, Dowdy E. Transcutaneous neuromuscular electrical stimulation (VitalStim) curative therapy for severe dysphagia: myth or reality? Ann Otol Rhinol Laryngol. 2007 Jan;116(1):36-44. doi: 10.1177/000348940711600107. PMID 17305276
- [Background] Logemann JA. The effects of VitalStim on clinical and research thinking in dysphagia. Dysphagia. 2007 Jan;22(1):11-2. doi: 10.1007/s00455-006-9039-2. Epub 2007 Jan 10. No abstract available. PMID 17216392
- [Background] Engelen MP, Orozco-Levi M, Deutz NE, Barreiro E, Hernandez N, Wouters EF, Gea J, Schols AM. Glutathione and glutamate levels in the diaphragm of patients with chronic obstructive pulmonary disease. Eur Respir J. 2004 Apr;23(4):545-51. doi: 10.1183/09031936.04.00022204. PMID 15083752
- [Background] Kargotich S, Keast D, Goodman C, Bhagat CI, Joske DJ, Dawson B, Morton AR. Monitoring 6 weeks of progressive endurance training with plasma glutamine. Int J Sports Med. 2007 Mar;28(3):211-6. doi: 10.1055/s-2006-924218. Epub 2006 Oct 6. PMID 17024635
- [Background] Holm E, Hack V, Tokus M, Breitkreutz R, Babylon A, Droge W. Linkage between postabsorptive amino acid release and glutamate uptake in skeletal muscle tissue of healthy young subjects, cancer patients, and the elderly. J Mol Med (Berl). 1997 Jun;75(6):454-61. doi: 10.1007/s001090050131. PMID 9231886
- [Background] Rutten EP, Franssen FM, Engelen MP, Wouters EF, Deutz NE, Schols AM. Greater whole-body myofibrillar protein breakdown in cachectic patients with chronic obstructive pulmonary disease. Am J Clin Nutr. 2006 Apr;83(4):829-34. doi: 10.1093/ajcn/83.4.829. PMID 16600935
- [Background] Fiatarone MA, O'Neill EF, Ryan ND, Clements KM, Solares GR, Nelson ME, Roberts SB, Kehayias JJ, Lipsitz LA, Evans WJ. Exercise training and nutritional supplementation for physical frailty in very elderly people. N Engl J Med. 1994 Jun 23;330(25):1769-75. doi: 10.1056/NEJM199406233302501. PMID 8190152
- [Background] Ouellette MM, LeBrasseur NK, Bean JF, Phillips E, Stein J, Frontera WR, Fielding RA. High-intensity resistance training improves muscle strength, self-reported function, and disability in long-term stroke survivors. Stroke. 2004 Jun;35(6):1404-9. doi: 10.1161/01.STR.0000127785.73065.34. Epub 2004 Apr 22. PMID 15105515
- [Background] Burgomaster KA, Hughes SC, Heigenhauser GJ, Bradwell SN, Gibala MJ. Six sessions of sprint interval training increases muscle oxidative potential and cycle endurance capacity in humans. J Appl Physiol (1985). 2005 Jun;98(6):1985-90. doi: 10.1152/japplphysiol.01095.2004. Epub 2005 Feb 10. PMID 15705728
- [Background] Weiner P, Magadle R, Berar-Yanay N, Davidovich A, Weiner M. The cumulative effect of long-acting bronchodilators, exercise, and inspiratory muscle training on the perception of dyspnea in patients with advanced COPD. Chest. 2000 Sep;118(3):672-8. doi: 10.1378/chest.118.3.672. PMID 10988188
- [Background] Gosselink R. Respiratory rehabilitation: improvement of short- and long-term outcome. Eur Respir J. 2002 Jul;20(1):4-5. doi: 10.1183/09031936.02.00402002. No abstract available. PMID 12166579
- [Background] Kim J, Sapienza CM. Implications of expiratory muscle strength training for rehabilitation of the elderly: Tutorial. J Rehabil Res Dev. 2005 Mar-Apr;42(2):211-24. doi: 10.1682/jrrd.2004.07.0077. PMID 15944886
- [Background] Sapienza CM, Davenport PW, Martin AD. Expiratory muscle training increases pressure support in high school band students. J Voice. 2002 Dec;16(4):495-501. doi: 10.1016/s0892-1997(02)00125-x. PMID 12512637